CLINICAL TRIAL: NCT04800120
Title: The Use of Hyperbaric Oxygen Therapy (HBOT) for the Treatment of COVID-19 Patients With Mild-to-moderate Respiratory Distress
Brief Title: Use of Hyperbaric Oxygen Therapy to Treat COVID-19 Patients With Respiratory Distress
Acronym: HBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB Protocol #00800
Record Dates: First submitted 2020-11-13; First posted 2021-03-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Study Group: Provide 100% oxygen at 2.0 ATA for 90 minutes on consecutive days for a total of up to 5 treatment to COVID-19 patients meeting inclusion criteria Control Group: Any COVID-19 positive patient meeting study inclusion criteria that does not receive HBOT (historical)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Identified COVID 19 patients receiving the intervention of Hyperbaric Oxygen Therapy
  Interventions: Other: Hyperbaric Oxygen Therapy
- Control Group (No Intervention): Historical control of COVID 19 patients who were previously treated and did not receiving Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — Delivery of 100% oxygen within a hyperbaric oxygen therapy chamber
  Other Names: HBOT
  Arms: Study Group

SUMMARY:
Investigate whether hyperbaric oxygen therapy treatment can become a viable treatment option for COVID-19. If successful, providers will be able to provide future COVID-19 patients with mild-to-moderate respiratory distress hyperbaric oxygen therapy in order to help avoid mechanical ventilation

DETAILED DESCRIPTION:
Using the Monoplace Hyperbaric Oxygen Chambers we will be providing COVID- 19 positive patients with mild-to-moderate distress 100% oxygen at 2.0 ATA for 90 minutes on consecutive days for a total of up to 5 treatments. A comparison will be made using a historical cohort not receiving HBOT. Data will be collected to determine whether or not HBOT is of any benefit to COVID-19 positive patient with mild-to-moderate respiratory distress.

Study Group: Provide 100% oxygen at 2.0 ATA for 90 minutes on consecutive days for a total of up to 5 treatment to COVID-19 patients meeting inclusion criteria Control Group: Any COVID-19 positive patient meeting study inclusion criteria that does not receive HBOT (historical) The control group is further defined as patients who were previously treated for COVID-19 at Morton Hospital that did not receive hyperbaric oxygen therapy. This will require accessing medical records to obtain patient information to establish the historical control data metric.

Study outcome measures:

* Time to normalize 02 requirement (ambient air pulse ox greater than or equal to 92% or ABG w/Pa02 greater than 60mmHG on air)
* Mortality
* Days free of invasive mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Verified COVID-19 infection
* Patient w/02 dependence of less than or equal to 6 liter/min to maintain pulse ox greater than or equal to 92% or arterial gas w/PA02 greater than 60mm HG

Exclusion Criteria:

* Not diagnosed w/COVID-19 infection
* Pregnancy
* DNR or other restrictions in escalation of level of care
* Contraindication for HBO
* Blood pressure parameters which are deemed unstable by clinical team
* Patients who require continuous ECG and/or continuous blood pressure monitoring, and with arterial lines
* Patients requiring rewarming
* Patients requiring any kind of invasive catheter/pressure monitoring
* Patients requiring continuous support of intravenous medication
* Minor subject (less than 18 years old)
* Refusal to participate
* Signs of respiratory decompensation requiring intubation and mechanical ventilation
* 02 dependence greater than or equal to 6L/minute to obtain Sa02 greater than or equal to 92% or ABG w/Pa02 >60mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Normalization of oxygen | through study completion, an average of 1 year
  normalize 02 requirement (ambient air pulse ox greater than or equal to 92% or ABG w/Pa02 greater than 60mmHG on air)

SECONDARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  Patient survival of COVID-19
Days free of invasive mechanical ventilation | through study completion, an average of 1 year
  The time which patient remains without the need for intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jill Trelease, DNP, Principal Investigator — Steward Healthcare
Locations (1):
- Morton Hospital, Taunton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No